CLINICAL TRIAL: NCT04725253
Title: Nicotinamide, an Inhibitor of PARP-1, for Preventing Delirium in Older Adults
Brief Title: Nicotinamide to Prevent Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, FONDECYT (Chile). (Unknown)
Responsible Party: Principal Investigator, Felipe Salech Morales, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FONDECYT 11190882
Record Dates: First submitted 2021-01-17; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Delirium Confusional State
MeSH Terms: conditions — Confusion | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: This randomized placebo-controlled trial.
Who Masked: Participant, Care Provider
Masking Description: The physician in charge will kept the randomization code, and no rater became aware of treatment allocations until requesting unmasking. Nurses were blinded except those who managed the study medication. All clinical staff, including nurses, physiotherapists or occupational therapist, will blinded. Patient and Family will be blind as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental): Patients who meet the inclusion / exclusion criteria will be randomly assigned to the experimental group:They will continue to receive standard prevention measures: Detection of delirium, education of health care team and the patient's family, sleep hygiene plan, early mobilization, resolve sensory impairments, and delivery of information of temporal-spatial reorientation in continuously. Study medication will be managed by nurses and administered daily at 7 a.m. This regimen will be continued up to 7 days after admission. The dosage of nicotinamide will be 1,5 gr per day.
  Interventions: Dietary Supplement: Nicotinamide
- Control (Placebo Comparator): Patients who meet the inclusion / exclusion criteria will be randomly assigned to the Control group: They will continue to receive the standard prevention measures: delirium detection, treatment health team education and the patient's family, sleep hygiene plan, early mobilization, resolve sensorial deterioration, and delivery of information of temporal-spatial reorientation in a continuous manner. Study medication will be managed by nurses and administered daily at 7 a.m. (in these case placebo tablets). This regimen will be continued up to 7 days after admission.
  Interventions: Other: Placebo tablets

INTERVENTIONS:
Dietary Supplement: Nicotinamide — Nicotinamide, 1,5 gr per day for 7 days.
  Arms: Nicotinamide
Other: Placebo tablets — Placebo tablets, 1 per day for 7 days.
  Arms: Control

SUMMARY:
Delirium is defined as an acute change in mental status characterized by fluctuating disturbances of consciousness, attention, cognition, and perception, usually secondary to acute injuries such as trauma or infections. Delirium is more frequent in older adults, and is associated with important poor clinical outcomes including increased mortality, functional deterioration, and higher expenditures for healthcare systems.

Although it is not the only one responsible, the inflammatory response plays a key role in the development of delirium. From the first descriptions of the condition 2500 years ago, it is known that patients who present with inflammatory injuries such as trauma (pe. hip fracture) or infections (sepsis), frequently develop delirium. Microglia, are an inflammatory cell with phagocytic capacity, that inhabit the nervous system and have a critical role in the regulation of the inflammatory response in the brain. It is known that microglia have receptors that respond to systemic inflammatory mediators by generating new inflammatory mediators that exert their effect on other glial cells and neurons in the central nervous system, affecting their function. Mouse models have shown that depleting the brain of microglia prevents cognitive decline after a traumatic bone injury, suggesting a role of these cells in the development of delirium.

Poly(ADP-ribose) polymerase-1 (PARP-1) is a nuclear enzyme that participates in DNA repair, and in the regulation of the expression of inflammatory mediators by immune cell. In vitro experiments have shown that PARP-1 enhances the microglial response to inflammation, and data from mice exposed to the bacterial component "lipo-poly-saccharide (LPS)", a classical model of delirium, showed that pharmacological inhibition of PARP-1 prevents cognitive decline secondary to that injury. Interestingly, nicotinamide, a vitamin widely available in the market, with a well-known safety profile in humans, is a well-recognized inhibitor of PARP-1. The role of PARP-1 nor nicotinamide in delirium has never been explored.

Considering that, 1) there is evidence showing that PARP-1 may act as an enhancer of the inflammatory response of microglia and 2) the protective effect against cognitive impairment produced by pharmacological inhibition of PARP-1 in a mice model of delirium, we propose as hypothesis that PARP-1 participates in delirium pathogenesis by enhancing microglial activation in response to systemic inflammation. To address this hypothesis in patients, we propose to determine in a randomized clinical trial whether nicotinamide, a pharmacological inhibitor of PARP-1, is more effective than placebo for the prevention of delirium in older adults with requirement of oxygen (non-invasive) and suspected coronavirus disease (COVID-19) under study.

The results of this research will contribute significantly in the field of delirium, improving the knowledge of its physiopathology, as well with the development of of new alternatives for its prevention in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Older than 65 years old.
* Newly admitted due to suspected coronavirus disease (COVID-19) under study.
* To have less than 24 hours from the hospitalization at the moment of randomization.
* Able to take medicine orally.
* Signed an informed consent.

Exclusion Criteria:

* An expected stay or life expectancy of less than 48 hours.
* Severe liver dysfunction or Lewy body disease.
* Syndromes associated with alcohol dependency and drug abuse.
* Psychotic or bipolar disorders receiving treatment with antipsychotics.
* Delirious at admission Patients.
* Documented viral infections.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-01-21 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium during the 1 week after injury. | 7 days
  The Confusion Assessment Method (CAM) will be used to measure delirium. CAM will be assessed between 10 and 11 a.m., and between 8 and 9 p.m. in all patients (twice a day for 7 days).

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Salech, MD PhD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No